CLINICAL TRIAL: NCT04666181
Title: Effects of Dual-Task Training on Cognitive and Motor Learning and Cortical Activation in Healthy Young Adults
Brief Title: Cortical Activation and Cognitive-Motor Learning
Acronym: Co-ACT&LEARN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Swati Manoharrao Surkar, Assistant Professor, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-001938
Record Dates: First submitted 2020-11-23; First posted 2020-12-14 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Dual-task; Healthy Adults
Keywords: Cognition; Motor; Dual-task; Prefrontal cortex; Sensorimotor cortex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual-task training (Experimental): Dual-task training will consist of balancing on the dynamic stability platform and responding to auditory stimuli. Participants will perform 18 trials total in 3 blocks of 6 trials. Each trial will be 30 seconds (s) in duration followed by 30 s of rest (i.e. quiet standing on the platform while holding onto the rails.) Between each training block, the participant will step off the platform and rest for 2 minutes. Dual-task training will occur on consecutive visits 2-6.
  Interventions: Behavioral: Dual-task training

INTERVENTIONS:
Behavioral: Dual-task training — See descriptions under arm description. The dual-task training will occur across a total of 5 consecutive workday visits.

SUMMARY:
The purpose of this research study is to assess the effects of dual-task training using a dynamic balance task and an auditory reaction time task on dual-task performance in healthy young adults and to assess the cortical activity within the prefrontal and sensorimotor cortices in response to dual-task training using functional near infrared spectroscopy (fNIRS).

DETAILED DESCRIPTION:
The purpose of this study is to assess the influence of a dual-task (combined motor-cognitive task) on dual-task performance of a complex dynamic stability task in healthy young adults and to assess the effects of dual-task training on cognitive-motor learning and cortical activation in healthy young adults. A dual-task is defined as concurrent performance of two tasks, usually a cognitive and motor task, that can be performed independently and have distinct and separate goals. Individuals engage in dual tasks every day and must allocate attentional resources to each task. While recognition of susceptibility to performance decrements in dual-task settings may be difficult, increased dual-task complexity is associated with decreased performance in one or both tasks. The well documented effects of dual-task practice represent a promising approach to improve dual-task performance for clinical populations such as individuals with neurological conditions or older individuals, in which complex multitask situations can increase fall risk due to hindered balance and walking performance. Similarly, young adults have demonstrated performance decrements while executing a dual-task that involved a combined balance and cognitive task. Research of dual-task training in healthy young cohort has indicated significant improvements in both motor and cognitive task performance in dual-task situations, suggesting the efficiency of this intervention strategy. However, most of these studies have investigated effects of a simple postural task combined with cognitive task training on dual-task performance. Effects of dual-task training using a complex dynamic postural stability task on dual-task performance of such complex task is lacking. Moreover, existing studies demonstrate conflicting evidence of dual-task training effects among healthy young adults since improvements in the motor task only have been largely reported. It is crucial to understand dual-task training effects on performance of a complex cognitive-motor task since postural control involves complex integration of somatosensory, vestibular, and visual systems. Our experimental paradigm will challenge these systems; thus, findings of this study would inform our intervention strategies in a variety of populations ranging from athletes to individuals with neurological conditions.

Dynamic postural stability is an integral aspect of postural control and it involves complex interaction of prefrontal, somatosensory, vestibular, and visual systems. However, a motor task involving complex interaction of these systems combined with cognitive task challenges has not been investigated thoroughly. Moreover, neural activation within these cortical areas during dual-task performance and effects of dual-task training are largely unknown.

Since, coordinated control of the body requires integration of all these systems (i.e. prefrontal, somatosensory, vestibular, and visual), it is important to systemically study the interference of an additional attention-demanding task, such as an auditory stimulus reaction time task on interaction of these systems that may contribute to decreased postural stability. Moreover, it is important to investigate if training on such a complex dual-task can reduce motor-cognitive interference, improve postural stability, and optimize cortical activation in complex dual-task conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy young adults
2. Right-handed

Exclusion Criteria:

1. Individuals with cognitive deficits or communication problems
2. Individuals with impaired vision
3. Individuals with balance disorders such as vestibular disorders, etc.
4. Individuals with known cardiorespiratory dysfunctions
5. Individuals with presence of lower extremity condition, injury, or surgery within last 3 months which could compromise training
6. Individuals with history of concussion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in auditory reaction time task performance | Baseline to 10 days, and upto 3 weeks. Shorter reaction time indicates better performance.
  Average amount of time in seconds for a button press in response to an auditory tone
Change in balance task performance | Baseline to 10 days, and upto 3 weeks
  The average amount of time in seconds that a participant maintains the stability platform within 3 degrees of horizontal position during 6 trials of 30 sec each. The total score will range between 0-30 s. Higher balance score indicates better balance performance.
Change in dual-task performance | Baseline to 10 days, and upto 3 weeks
  Dual-task performance will assess performance on the combined auditory reaction time task and the balance task, i.e. performance under influence of dual-task situation.
Change in Cortical Activation | Baseline to 10 days, and upto 3 weeks
  The amount of change in cortical activity (change in oxyhemoglobin concentration in umol) within the prefrontal and sensorimotor cortices in response to dual-task training.

SECONDARY OUTCOMES:
Errors in auditory reaction time task performance | Baseline to 10 days, and upto 3 weeks
  Error is a wrong button pressed in response to the auditory tone
Balance variability | Baseline to 10 days, and upto 3 weeks
  The average amount of time in seconds on the left and right side of the dynamic stability platform outside of 3 degrees in the center during 6 trials of 30 seconds each. Smaller time on the right and left side indicates improvement in variability.

CONTACTS AND LOCATIONS:
Overall Officials: Swati M Surkar, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will share after the completion of the study upon request to the PI.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available immediately after completion of the study.

REFERENCES:
- [Background] Beauchet O, Dubost V, Herrmann FR, Kressig RW. Stride-to-stride variability while backward counting among healthy young adults. J Neuroeng Rehabil. 2005 Aug 11;2:26. doi: 10.1186/1743-0003-2-26. PMID 16095533
- [Background] Fraser SA, Li KZ, Berryman N, Desjardins-Crepeau L, Lussier M, Vadaga K, Lehr L, Minh Vu TT, Bosquet L, Bherer L. Does Combined Physical and Cognitive Training Improve Dual-Task Balance and Gait Outcomes in Sedentary Older Adults? Front Hum Neurosci. 2017 Jan 18;10:688. doi: 10.3389/fnhum.2016.00688. eCollection 2016. PMID 28149274
- [Background] Ghai S, Ghai I, Effenberg AO. Effects of dual tasks and dual-task training on postural stability: a systematic review and meta-analysis. Clin Interv Aging. 2017 Mar 23;12:557-577. doi: 10.2147/CIA.S125201. eCollection 2017. PMID 28356727
- [Background] Kiss R, Brueckner D, Muehlbauer T. Effects of Single Compared to Dual Task Practice on Learning a Dynamic Balance Task in Young Adults. Front Psychol. 2018 Mar 12;9:311. doi: 10.3389/fpsyg.2018.00311. eCollection 2018. PMID 29593614
- [Background] Pinti P, Tachtsidis I, Hamilton A, Hirsch J, Aichelburg C, Gilbert S, Burgess PW. The present and future use of functional near-infrared spectroscopy (fNIRS) for cognitive neuroscience. Ann N Y Acad Sci. 2020 Mar;1464(1):5-29. doi: 10.1111/nyas.13948. Epub 2018 Aug 7. PMID 30085354
- [Background] Techayusukcharoen R, Iida S, Aoki C. Observing brain function via functional near-infrared spectroscopy during cognitive program training (dual task) in young people. J Phys Ther Sci. 2019 Jul;31(7):550-555. doi: 10.1589/jpts.31.550. Epub 2019 Jul 9. PMID 31417220

DOCUMENTS (1):
  • Informed Consent Form (2020-09-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT04666181/ICF_000.pdf